CLINICAL TRIAL: NCT00001035
Title: A Phase I Pilot Study of the Safety and Efficacy of Interferon Alfa-2b (IFN Alfa-2b) in Combination With Nucleoside Analog Therapy in Patients With Combined Hepatitis C (HCV) and Advanced Human Immunodeficiency Virus (HIV) Infections
Brief Title: The Safety and Effectiveness of a Two-Drug Combination in the Treatment of Patients With Hepatitis C Plus Advanced HIV Infections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 203P; 11180 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: HIV Infections; Hepatitis C
Keywords: AIDS-Related Opportunistic Infections; Interferon Alfa-2b; Zalcitabine; Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Zidovudine; Hepatitis C
MeSH Terms: conditions — HIV Infections; Hepatitis C; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Interferon alpha-2; Zidovudine; Zalcitabine; Didanosine

INTERVENTIONS:
Drug: Interferon alfa-2b
Drug: Zidovudine
Drug: Zalcitabine
Drug: Didanosine

SUMMARY:
To investigate the toxicity of interferon alfa-2b ( IFN alfa-2b ) in combination with nucleoside analog therapy in HIV-positive patients with chronic hepatitis C. To determine the efficacy of treatment with IFN alfa-2b for chronic hepatitis C in patients with advanced HIV infections treated with nucleoside analog therapy.

IFN alfa-2b has HIV inhibitory properties and has also been approved for treatment of chronic hepatitis C. Studies have shown that IFN alfa-2b is effective in asymptomatic HIV-positive patients with chronic hepatitis C, but the drug's benefit against hepatitis C in patients with advanced HIV infection has not been determined.

DETAILED DESCRIPTION:
IFN alfa-2b has HIV inhibitory properties and has also been approved for treatment of chronic hepatitis C. Studies have shown that IFN alfa-2b is effective in asymptomatic HIV-positive patients with chronic hepatitis C, but the drug's benefit against hepatitis C in patients with advanced HIV infection has not been determined.

Patients receive interferon alpha-2b subcutaneously 3 times weekly for 6 months. If no response is seen after 18 weeks of therapy or if an initial response is followed by relapse while on therapy, dose is increased. Patients who require a dose escalation should continue on IFN alfa-2b for an additional 6 months. All patients will also receive available nucleoside analog therapy ( zidovudine, didanosine, zalcitabine ) at currently accepted doses as clinically appropriate.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Treatment or suppression of opportunistic infections with standard drugs.
* Pneumovax, HIB, tetanus, influenza, and hepatitis B vaccines.
* Clinically indicated antibiotics.
* Short courses of steroids (< 21 days) for acute problems not related to hepatitis C.
* Other regularly prescribed medications such as analgesics, nonsteroidal anti-inflammatory agents, antipyretics, allergy medications, and oral contraceptives.

Patients must have:

* HIV positivity.
* Documented hepatitis C virus.
* CD4 count <= 200 cells/mm3.
* No severe liver disease (Grade C Childs-Pugh classification) or chronic liver disease not caused by hepatitis C.
* Willingness to be followed for the duration of treatment and follow-up period.

Prior Medication:

Allowed:

* Prior AZT, ddI, and ddC.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Hepatitis B (HBsAg positive).
* Autoimmune hepatitis (FANA titer >= 1:160 and anti-smooth muscle antibody titer >= 1:160).
* Wilson's disease.
* alpha-1 antitrypsin deficiency.
* Hemochromatosis.
* Malignancy requiring systemic chemotherapy.

Concurrent Medication:

Excluded:

* Nonnucleoside analog therapy for HIV.
* Biologic response modifiers.
* Systemic cytotoxic chemotherapy.
* Chronic systemic steroid use.

Concurrent Treatment:

Excluded:

* Radiation therapy other than local irradiation to the skin.

Prior Medication:

Excluded:

* Prednisone within 12 weeks prior to study entry (if patient has received prior daily doses for 1 month or longer duration).
* Acute therapy for an infection within 2 weeks prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gill JC, Study Chair; Eyster ME, Study Chair
Locations (3):
- United States (3):
  - USC CRS, Los Angeles, California
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - NY Univ. HIV/AIDS CRS, New York, New York